CLINICAL TRIAL: NCT00407329
Title: Urokinase Plasminogen Activator System in Benign Prostatic Hyperplasia: A Possible Marker of Progression and Response to Medical Therapy
Brief Title: Urokinase Plasminogen Activator System in Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. J. Curtis Nickel, Professor, Queen's University
Other Study IDs: uPAR
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: BPH
Keywords: BPH
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: transurethral resection of the prostate — resection of prostate
  Other Names: TURP

SUMMARY:
We hypothesize that the absolute or relative serum or urine levels of the urokinase plasminogen activator system, including uPA, uPAR and PAI-1,2 (inhibitors of the uPAR/uPA complex), are associated with inflammation in prostatic tissue.

DETAILED DESCRIPTION:
Histological inflammation in patients with Benign Prostatic Hyperplasia (BPH) appears to predict clinical progression and ultimate long-term response to various medical therapies, including finasteride. Discovery of a urine or serum marker of prostate inflammation will be an invaluable clinical tool to predict a man's risk of BPH progression and the efficacy of various medical therapies to reduce that risk.

Specific Aim:

We plan to determine if urokinase plasminogen activators (and/or other inflammatory markers) in serum, urine and tissue of patients can predict prostatic inflammation

Background:

Benign Prostatic Hyperplasia (BPH) and Inflammation

BPH is a common disorder of the prostate causing significant lower urinary tract symptoms and negatively affects the quality of life in a substantial proportion of men in North America. According to the National Institutes of Health (NIH), BPH affects more than 50% of men over age 60 and as many as 90% of men over the age of 70. Although there are numerous genetic and epigenetic changes associated with the progression of normal prostatic glandular formation to BPH, as early as 1994 our group suggested that the presence of prostatic inflammation could be associated with pathogenesis and progression of both histological and clinical BPH. We have demonstrated that histological prostate inflammation is very common in patients with BPH as well as patients who are both symptomatic and not symptomatic. Our local research group spearheaded an international consensus classification system for prostatic inflammation that we have subsequently employed in our ongoing study of over 8,000 men undergoing 3 serial biopsies over a 4 year period of time. The MTOPS BPH study data base subanalyses of the more than 1,000 men who underwent baseline biopsies strongly suggested that prostatic inflammation appears to be the strongest and most robust predictor of symptomatic progression as well as response to drug therapy. An analyses T-cell phenotypes, cytokine expression patterns and cellular cross talk in BPH tissues of 101 BPH patients and prostatic cell cultures showed that chronic inflammation triggers histological and clinical progression. The search for urine or serum biomarkers of prostatic inflammation is highly relevant to better target therapies for men with this common condition.

Urokinase Plasminogen Activator System

Proteolytic enzymes are required to mediate inflammatory cell infiltration in tissues, a process highly regulated by the cell surface-specific receptor (uPAR) a binding partner for the urokinase-type plasminogen activator (uPA). Numerous previous clinical investigations have indicated that serum levels of the plasminogen activation system are an effective marker of inflammation in several disease processes including CNS inflammation, asthma, metabolic syndrome and pre-eclampsia. Very little data is available regarding the plasma levels of soluble uPAR in benign prostatic diseases, although one previous report suggested higher average levels of soluble uPAR in patients with lower urinary tract symptoms. Theses authors reported a wide variation of uPAR in BPH patients with some having greatly elevated levels while others had undetectable levels. However, the author's did not have pathological confirmation of their findings and could not quantify the level of inflammation in the prostatic tissue. We hypothesize that the absolute or relative serum levels of the urokinase plasminogen activator system, including uPA, uPAR and PAI-1,2 (inhibitors of the uPAR/uPA complex), are associated with inflammation in prostatic tissue.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for transurethral resection of the prostate

Exclusion Criteria:

* unable to give consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men needing TURP
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Curtis Nickel, MD FRCSC, Principal Investigator — Queen's Universtiy
Locations (1):
- Centre for Advanced Urological Research, Kingston, Ontario, Canada

REFERENCES:
- [Background] Nickel JC. Prostatic inflammation in benign prostatic hyperplasia - the third component? Can J Urol. 1994 Jan;1(1):1-4. PMID 12834558
- [Background] Nickel JC, Downey J, Young I, Boag S. Asymptomatic inflammation and/or infection in benign prostatic hyperplasia. BJU Int. 1999 Dec;84(9):976-81. doi: 10.1046/j.1464-410x.1999.00352.x. PMID 10571623
- [Background] Nickel JC, True LD, Krieger JN, Berger RE, Boag AH, Young ID. Consensus development of a histopathological classification system for chronic prostatic inflammation. BJU Int. 2001 Jun;87(9):797-805. doi: 10.1046/j.1464-410x.2001.02193.x. PMID 11412216
- [Background] McCabe NP, Angwafo FF 3rd, Zaher A, Selman SH, Kouinche A, Jankun J. Expression of soluble urokinase plasminogen activator receptor may be related to outcome in prostate cancer patients. Oncol Rep. 2000 Jul-Aug;7(4):879-82. doi: 10.3892/or.7.4.879. PMID 10854562
- [Background] McConnell JD, Roehrborn CG, Bautista OM, Andriole GL Jr, Dixon CM, Kusek JW, Lepor H, McVary KT, Nyberg LM Jr, Clarke HS, Crawford ED, Diokno A, Foley JP, Foster HE, Jacobs SC, Kaplan SA, Kreder KJ, Lieber MM, Lucia MS, Miller GJ, Menon M, Milam DF, Ramsdell JW, Schenkman NS, Slawin KM, Smith JA; Medical Therapy of Prostatic Symptoms (MTOPS) Research Group. The long-term effect of doxazosin, finasteride, and combination therapy on the clinical progression of benign prostatic hyperplasia. N Engl J Med. 2003 Dec 18;349(25):2387-98. doi: 10.1056/NEJMoa030656. PMID 14681504
- [Background] Thompson IN, Goodman PJ, Tangen CM, Lucia MS, Miller CJ, Ford LC, et al. The influence of finsteride in the development of prostate cancer. New England Journal of Medicine, 2003; 349:211-220.